CLINICAL TRIAL: NCT02485600
Title: Canadian Advanced Parkinson DUODOPA-Treated Patients Observational Study Evaluating Long-Term Health Outcomes in Centers of Excellence (CADENCE)
Brief Title: Observational Study Evaluating Long-term Health Outcomes of Canadian DUODOPA-treated Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-506
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease (PD)
Keywords: Cadence; Duodopa; Parkinson's disease; LCIG; Levodopa-carbidopa intestinal gel; Observational
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DUODOPA patients.: Patients starting DUODOPA treatment at time of enrollment.

SUMMARY:
This is an open-label, postmarketing, observational study to document health outcomes, in Canadian patients with advanced Parkinson's disease and long-term treatment with Duodopa (levodopa/carbidopa intestinal gel).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced Parkinson's Disease
* Prescribed Duodopa by his/her treating physician.

Exclusion Criteria:

* Patients who were previously treated with Duodopa.
* Presence of other condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of advanced PD.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of patients eligible for DUODOPA treatment according to the DUODOPA Product Monograph (DPM) approved by Health Canada and according to the reimbursement criteria accepted by the Canadian Provincial Health Authorities or private insurance companies.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in participant's motor symptoms | Baseline, Day 1, Month 3, Month 6, and every 6 months thereafter up to 48 months
  Evaluated via the Unified Parkinson's Disease Rating Scale (UPDRS) Part II, III, V and Part IV items 33-35; items 32 & 39 modified as per MDS-UPDRS, and the Freezing of Gait Questionnaire (FOGQ).
Change in the cognitive functions. | Baseline, Day 1, and every 12 months thereafter up to 48 months
  Evaluated via the Montreal Cognitive Assessment (MoCa).
Change in the Parkinson's Disease Questionnaire (PDQ-39) | Baseline, Day 1, Month 3, and every 6 months thereafter up to 48 months
  Evaluated via the Parkinson's Disease Questionnaire (PDQ-39)
Change in caregiver burden | Baseline, Day 1, Month 3, and every 6 months thereafter up to 48 months
  Evaluated via the Zarit Care Giver Burden Questionnaire.
Change in the non-motor symptoms. | Baseline, Day 1, Month 3, and very 6 months thereafter up to 48 months
  Evaluated via the Non-Motor symptoms Scale (NMS) and the Parkinson's Disease Sleep Scale (PDSS-2).
Change in caregiver work productivity | Baseline, Day 1, Month 3, and every 6 months thereafter up to 48 months
  Evaluated by the Work Productivity and Activity Information Questionnaire (WPAI - care giver)
Change in the participant's Healthcare Resource Utilization | Baseline, Month 3, and every 6 months thereafter up to 48 months
  Evaluated via the Health Care Resources Utilization Questionnaire (HCRU).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (13):
- Canada (13):
  - University of Calgary /ID# 151948, Calgary, Alberta
  - Zeidler Ledcor Centre /ID# 135979, Edmonton, Alberta
  - St. Boniface Clinic, CA /ID# 162092, Winnipeg, Manitoba
  - Hamilton Health Sciences /ID# 148808, Hamilton, Ontario
  - Kingston General Hospital /ID# 144942, Kingston, Ontario
  - London Health Sciences Centre /ID# 138434, London, Ontario
  - The Ottawa Hospital /ID# 135981, Ottawa, Ontario
  - Toronto Western Hospital /ID# 135980, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 135977, Montreal, Quebec
  - McGill Univ HC /ID# 138334, Montreal, Quebec
  - Ctr Hosp Enfant Jesus /ID# 138435, Québec, Quebec
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 144941, Québec, Quebec
  - CHUS - Hopital Fleurimont /ID# 148811, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/levodopa_carbidopa_P14-506.pdf